CLINICAL TRIAL: NCT01314859
Title: ADMINISTRATION OF NIFIDEPINE VERSUS ATOSIBAN IN PREGNANT WOMEN WITH A THREAT OF PREMATURE LABOR
Brief Title: Nifedipine Treatment in Preterm Labor
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Fundación Ramón Domínguez (Other)
Responsible Party: Manuel Macía Cortiñas, MD, Hospital Clínico de Santiago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC-NIF-2010-01; 2010-024122-37 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2011-02

CONDITIONS: Threatened Preterm Labor
Keywords: Nifedipine; Obstetric Labor; Premature; Tocolysis
MeSH Terms: conditions — Premature Birth | interventions — Nifedipine; atosiban

ARMS (2):
- Nifedipine (Experimental): * Oral Treatment with Nifedipine capsules (10 mg)
    * Initial dose: 20 mg of nifedipine (2 capsules of 10 mg).
    * Maintenance Dose: 20 mg of nifedipine (2 capsules of 10 mg) every 6 hours.
  * Maximum Duration of the treatment: 48 hours.
  Interventions: Drug: Nifedipine
- Atosiban (Active Comparator): * Intravenously Treatment with Atosiban (7.5mg/ml)
    * Initial Dose: IV bolus injection during 1 minute + Intravenous infusion 7.5 mg/ml during 3 hours.
    * Maintenance: Maintenance intravenous infusion 7.5 mg/ml at least 18 hours to a maximum of 45 hours.
  * Maximum Duration of the treatment: 48 hours.
  Interventions: Drug: Atosiban

INTERVENTIONS:
Drug: Nifedipine — * Oral Treatment with Nifedipine capsules (10mg)
    * Initial dose: 20 mg of nifedipine (2 capsules of 10 mg).
    * Maintenance Dose: 20 mg of nifedipine (2 capsules of 10 mg) every 6 hours.
  * Maximum Duration of the treatment: 48 hours.
  Arms: Nifedipine
Drug: Atosiban — * Intravenously Treatment with Atosiban (7.5mg/ml)
    * Initial Dose: IV bolus injection during 1 minute + Intravenous infusion 7.5 mg/ml during 3 hours.
    * Maintenance: Maintenance intravenous infusion 7.5 mg/ml at least 18 hours to a maximum of 45 hours.
  * Maximum Duration of the treatment: 48 hours.
  Arms: Atosiban

SUMMARY:
This is a study for pregnant women who have been diagnosed with Threatened Preterm Labor. The principal aim of this study is to compare the efficacy and safety of Nifedipine treatment versus Atosiban treatment over these patients' newborn babies.

DETAILED DESCRIPTION:
Preterm labor is defined as the presence of uterine contractions of sufficient frequency and intensity to effect progressive effacement and dilation of the cervix prior to term gestation (between 20 and 37 weeks).

It is a major health problem of increased incidence, affecting approximately between 7-10% of pregnant women in developed countries with a high socioeconomic costs and high rates of fetal mortality, although perinatal progress.

This study may allow to establish the existence of differences in perinatal outcomes and to define the first choice drug for tocolysis.

ELIGIBILITY:
Inclusion Criteria:

The study population and the inclusion criteria is established by patients between the 24th and 33+6th weeks of pregnancy, fixed by an ecography during the first three-month period, and with a threat of preterm labor (TLP), by the American College of Obstetricians and Gynecologists (ACOG's) criteria:

* Four contractions or more with a duration of at least 30 seconds during 30 minutes
* Documented cervix changes:

  * The cervix changes in a nulliparous woman are: both cervix tact with 0 to 4 cm of dilatation and cervical effacement of at least a 50% (vaginal ultrasound alternative with cervix length two standard curvatures under the average for the gestational age)
  * The cervix changes in a multiparous woman are: 1 to 4 cm of dilatation and cervical effacement of at least a 50% (same ecographic alternative as the nulliparous).
* Patient who had signed the informed consent.

Exclusion Criteria:

Exclusion criteria of the pregnant mother and intrauterine fetal:

* Prior treatment with a different tocolytic from the ones in the protocol.
* Chorioamnionitis.
* Premature rupture of membranes.
* Vaginal Bleeding.
* Major fetal malformations.
* Intrauterine growth retardation (IGR): IGR<percentile 5.
* Cardiopathies (aortic stenosis, congestive heart failure).
* Blood Pressure lower than 100/60 mmHg.
* High transaminase levels.
* Uterine malformations.
* Use of magnesium sulphate.
* Severe hypertensive disorder, defined as blood pressure equal to or greater than 160/100 mmHg or any figure associated with severe preeclampsia.
* Non-reassuring cardiac frequency tracing defined as category II and III of National Institute of Child Health and Human Development (NICHD).
* Asthmatic patients treated with betamimetics.
* Hypertensive patients treated with vasodilators.
* Patient in treatment or treated with another product/s in investigation during the four weeks prior to randomization.
* Hypersensitivity to any drug of the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Neonatal Respiratory Distress Syndrome (RDS) at birth | Measured in the newborn at birth and at 30 days after labor
  * Clinical assessment: results of the Silverman test. Existence of tachypnea, chest wall retractions, auricular flutter, expiratory grunting and chest-abdominal asynchrony.
  * Need of 02 at birth (maximum Fi02 in the first 24 hours to estimate the immediate distress). Measurement of pCO2 at birth.
  * Need of mechanic ventilation: invasive/not invasive and duration of it.
  * Radiologic estimation of the level of hyaline membrane disease
  * Need of a surfactant and number of used dosages.

SECONDARY OUTCOMES:
Prolongation of the pregnancy in women with Threatened Preterm Labor | more than 48 hours/7 days
  It will be evaluated as a delay in the labor: hours after starting the treatment: more than 48 hours/more than 7 days of prolongation.
Obstetric results | at labor and 24 hours after delivery
  Number of days and type of labor.
Presence of the neonatal intracranial hemorrhage | First assessment: in the first week.
  Determination of the appearance and periventricular hemorrhage degree (I-IV) by transfontelar ultrasound scans.
Presence of neonatal necrotizing enterocolitis | at birth and at 30 days after labor
  Monitor the need of canalizing the umbilical vein or artery, the days of parenteral nutrition, days to the start of enteral nutrition, type of enteral nutrition (from the mother, artificial or mixed), start of the elimination of meconium, clinical data from the neonatal necrotizing enterocolitis(abdominal strain, vomiting, blood in the feces, septic appearance) and radiologic/ecographic (dilated bowel loops, intestinal pneumatosis, air in portal, pneumoperitoneum).
Presence of Retinopathy of prematurity (ROP) | Between the 4th and 6th week of baby life.
  Monitor the iGF1 (Insulin-like growth factor 1) levels on the 3rd week of life as well as an assessing the development of retinopathy.
Presence of ductus | At birth and 30 days after labor
  Clinical assessment (heart murmur, jumpy pulse, worsening of the clinical basal situation), echocardiography (confirmation of the ductus, Al/Ao relation, ductal size), medical or surgical treatment necessity.
Mother Tolerance Results | at labor and 24 hours after delivery
  Survey to assess the tolerance to the symptomatology induced by the medicines (flush, tachycardia, digestive upsets).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Macía Cortiñas, MD, Study Chair — Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain; Lourdes González González, MD, Principal Investigator — Hospital Son Dureta, Mallorca, Spain; Javier Martínez Pérez-Mendaña, MD, PhD, Principal Investigator — Complexo Hospitalario Arquitecto Marcide- Profesor Novoa Santos, Ferrol, Spain; José Eloy Moral Santamarina, MD, Principal Investigator — Complexo Hospitalario de Pontevedra, Pontevedra, Spain; Susana Blanco Pérez, MD, Principal Investigator — Complexo Hospitalario de Ourense; Ourense, Spain; Luis Miguel González Seijas, MD, Principal Investigator — Hospital del Barbanza; Ribeira, A Coruna, Spain; Emilio Cabo Silva, MD, Principal Investigator — Hospital del Salnes; Vilagarcía de Arousa, Pontevedra, Spain

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046